CLINICAL TRIAL: NCT06707272
Title: A Study of the Correlation Between Donor UDP-Glc and Transplanted Kidney Function
Status: Completed | Type: Observational
Sponsor: Qianghua Leng (Other)
Responsible Party: Sponsor-Investigator, Qianghua Leng, Principal Investigator, Third Affiliated Hospital, Sun Yat-Sen University
Organization: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Other Study IDs: II2024-047-02
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Renal Transplant
Keywords: renal transplant; delayed graft function; acute kidney injury
MeSH Terms: conditions — Delayed Graft Function; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — donors' blood samples and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- delayed graft function: Delay graft function (DGF) was defined as the need for dialysis treatment within the first week following transplantation or Scr at post-transplant 1 week (POW1) ≥ 4.52 mg/dL.
- Immediate graft function: Immediate graft function (IGF) was defined as Scr at POW1 < 2.50 mg/dL, and slow graft function (SGF) was defined as Scr at POW1 ≥ 2.50 mg/dL.

SUMMARY:
Kidney transplantation is the preferred treatment for end-stage renal disease (ESRD), however, organ shortage is the primary bottleneck restricting the progression of organ transplantation.1 Organs from Expanded Criteria Donors (ECD) have the potential to greatly increase the donor organ pool. However, they also require careful selection and utilization. Deceased kidney donors often had a history of central nervous system fluid regulation disorders and inflammation mediator release, which led to hemodynamic instability, electrolyte and acid-base imbalances, and with a higher risk of primary graft non-function (PNF) or delayed graft function (DGF) post-transplantation.2,3 Searching for appropriate and effective biomarkers to assess renal quality and predict DGF is a hot topic in the field of kidney transplantation.

Uridine diphosphate-glucose (UDP-Glc) is a damage-associated molecular pattern molecule (DAMPs) released by damaged cells.4 UDP-Glc is synthesized in the cytoplasm, then transported into the lumen of the endoplasmic reticulum and Golgi apparatus, where it regulates the synthesis of carbohydrates and acts as a substrate to facilitate glycosylation reactions.5 And UDP-Glc is an endogenous excitant of the G protein-coupled P2Y14 receptor.6 Additionally, the human P2Y14 receptor is expressed at high levels in adipose tissue, stomach, intestines, specific regions of the brain, skeletal muscle, spleen, lungs, and heart.7 UDP-Glc released plays a significant role in extracellular signaling within these tissues.8 Activation of P2Y14 promotes neutrophil infiltration, the recruitment of monocytes and macrophages, and the activation of the immune response, ultimately leading to tissue damage.9 Research has discovered that intercalated cells (ICs) in the collecting duct of the kidney act as sensors for UDP-Glc, and when the P2Y14 receptor on their apical membrane is activated, ICs produce chemotactic cytokines that attract neutrophils to the kidney, causing kidney inflammation and the onset of acute kidney injury (AKI).10,11 Furthermore, studies have shown that the concentration of UDP-Glc in the urine of AKI patients is higher compared to patients without AKI.12 UDP-Glc hydrolyzes slowly in the extracellular environment, which results in UDP-Glc being highly stable and easily detectable.5,13 In conclusion, donor urinary UDP-Glc can be serve as an appropriate and effective biomarkers to assess renal quality and predict DGF.

The study aimed to investigated the correlation between donor urinary UDP-Glc levels and graft function post-transplant in recipients. We hypothesized that the higher the donor urinary UDP-Glc levels, the more severe the kidney damage, resulting in a higher probability of DGF. It will provide transplant surgeons with a novel strategy to predict DGF earlier and more accurately without invasive procedures, while also reducing medical costs.

ELIGIBILITY:
Inclusion Criteria:

* donors who met the criteria for kidney donation
* recipients who met the criteria for kidney transplantation
* informed consent form signed
* organs from deceased donors
* completed the family consent form for human organ donation.

Exclusion Criteria:

* donors without urine samples
* recipients with multiple organ transplantation
* participation in other clinical trials
* recipients died in perioperation period
* recipients experienced kidney transplant nephrectomy in perioperation period
* recipients did not have a follow-up visit at our center with 1 month after being first discharged
* other features considered unsuitable by researchers.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This a single-center observational clinical study included recipients who underwent successful kidney transplantation and had donor urine samples at our center between June 2023 and August 2024.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Post-transplant renal function | Within 7 days of kidney transplantation
  Assessment of patients' renal function recovery by serum creatinine values after renal transplantation

SECONDARY OUTCOMES:
Survival time of transplanted kidneys | Within 1 year after kidney transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Raw and post-statistical data
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: Upon completion of the clinical study and related publications
Access Criteria: Anyone wishing to access the data will be able to contact the corresponding author by email for access to the raw data.

REFERENCES:
- [Derived] Ma M, Han F, Leng Q, Chen X, Tang Z, Zhang J, Luo Y, Zhang Y, Huang Z, Na N. Preoperative donor urinary UDP-Glc as an independent risk factor for delayed graft function. Front Immunol. 2025 Mar 17;16:1545280. doi: 10.3389/fimmu.2025.1545280. eCollection 2025. PMID 40165952